CLINICAL TRIAL: NCT06671392
Title: A Multi-center, Randomized, Double-blind, Parallel Design, Phase III Study to Evaluate and Compare the Efficacy and Safety of DWC202405/DWC202313 and DWC202314 Combination Therapy to DWC202405/DWC202313 in Patients With Essential Hypertension Inadequately Controlled With DWC202405
Brief Title: A Phase III Study to Efficacy and Safety of DWC202405/DWC202313 and DWC202314 in Patients With Hypertension
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW_DWJ1622301
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DWC202405 (Experimental)
  Interventions: Drug: DWC202405
- DWC202405, DWC202314 / DWC202313, DWC202314 (Experimental)
  Interventions: Drug: DWC202405, DWC202314; Drug: DWC202313, DWC202314
- DWC202405, DWC202314P / DWC202313, DWC202314P (Placebo Comparator)
  Interventions: Drug: DWC202405, DWC202314P; Drug: DWC202313, DWC202314P

INTERVENTIONS:
Drug: DWC202405 — 5/20mg, 1 tablet, Oral, Once a day
  Arms: DWC202405
Drug: DWC202405, DWC202314 — 5/20mg + 1.5mg, 1 tablet, Oral, Once a day
  Arms: DWC202405, DWC202314 / DWC202313, DWC202314
Drug: DWC202405, DWC202314P — 5/20mg + 1.5mg, 1 tablet, Oral, Once a day
  Arms: DWC202405, DWC202314P / DWC202313, DWC202314P
Drug: DWC202313, DWC202314 — 10/40mg + 1.5mg, 1 tablet, Oral, Once a day
  Arms: DWC202405, DWC202314 / DWC202313, DWC202314
Drug: DWC202313, DWC202314P — 10/40mg + 1.5mg, 1 tablet, Oral, Once a day
  Arms: DWC202405, DWC202314P / DWC202313, DWC202314P

SUMMARY:
A Multi-center, Randomized, Double-blind, Parallel design, Phase III study to Evaluate and Compare the Efficacy and Safety of DWC202405/DWC202313 and DWC202314 Combination Therapy to DWC202405/DWC202313 in Patients with Essential Hypertension Inadequately Controlled with DWC202405

ELIGIBILITY:
Inclusion Criteria:

* Average systolic blood pressure (MSSBP) and average diastolic blood pressure (MSDBP) measured at the time of screening meet the following criteria (a) If antihypertensive drugs are being administered: 140 mmHg ≤ MSSBP < 180 mmHg and MSDBP < 110 mmHg However, the criteria of 130 mmHg ≤ MSSBP < 180 mmHg and MSDBP < 110 mmHg are applied to patients with the following diseases.

Exclusion Criteria:

* If the blood pressure measured at the time of screening and randomization is MSSBP ≥ 180 mmHg or MSDBP ≥ 110 mmHg
* Those whose blood pressure differences measured on both arms at the time of screening are MSSBP ≥ 20 mmHg and MSDBP ≥ 10 mmHg

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
change of MSSBP (Mean Sitting Systolic Blood Pressure) based on baseline | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University ANAM Hospital, Seoul, South Korea